CLINICAL TRIAL: NCT01428323
Title: Study of the Aerosol Deposition With Vented and Unvented Jet Nebulizer in Healthy Subjets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 3.4529.10
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Aerosol Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vented and Unvented Jet Nebulizer — Nebulizers used with 500mg aminoglycosides in 4ml until One minute after the sputerring point.
  Other Names: Nebulizer Type: Sidestream

SUMMARY:
Open-vent jet nebulizers are frequently used to promote drug lung deposition but their clinical efficacy and indications are not clear.

Our study aimed to compare inhaled mass, and lung deposition of amikacin by using a jet nebulizer (Sidestream) under two different configurations: vented and unvented coupled to a 110 ml corrugated piece of tubing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers between 18 and 60 years old

Exclusion Criteria:

* Smokers
* Pathological spirometry
* History of treatment with aminoglygosides 1 month prior the study
* Known allergy to aminoglycosydes
* Any lung pathology or history of lung surgery

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Amikacin Urinatory excretion | Each miction during 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital, Belgium